CLINICAL TRIAL: NCT07018089
Title: The Efficacy of the iWork.COMP Among Health Care Professionals: A Randomized Controlled Trial
Brief Title: The Efficacy of the iWork.COMP Among Health Care Professionals
Acronym: iWorkCOMP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Collaborators: European Union (Horizon Europe Programme) (Unknown)
Responsible Party: Principal Investigator, Diana Ribeiro da Silva, Principal Investigator, University of Coimbra
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 101137244; HORIZON-HLTH-2023-CARE-04 (Other Grant/Funding Number: European consortium - KEEPCARING)
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Toxic Leadership Styles
Keywords: Health care workers; Surgical pathway; Clinical Trial; Compassion Focused Therapy; iWork.COMP
MeSH Terms: interventions — Health Personnel

STUDY DESIGN:
Intervention Model Description: This project will use a longitudinal design. The healthcare units will be randomly assigned to two conditions: the TG and WLCG. Considering that concealment of group allocation is not possible within the iWork.COMP (which is a transversal issue in any psycho-educative/psychotherapeutic approach), this specific RCT will not have a blinded design.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): The TG will receive iWork.COMP. The iWork.COMP is an 8-week internet delivery intervention based on CFT, aimed at reducing the impact of toxic leadership styles through the development of a compassionate motivation. After this period, participants will have access to the SOS-Button tool. Participants in this group will be assessed in four assessment-points (4-weeks intervals; approximately 10 minutes per assessment point): baseline, middle of the intervention, post-treatment, four-week follow-up.
  Interventions: Behavioral: iWork.Comp
- Waiting List Control Group (No Intervention): This group will not receive any intervention during the study period. However, the access to the iWork.COMP program (and then to the SOS-Button tool) will be available after the study completion, if they choose to. Participants in this group will be assessed in four assessment-point (4-weeks intervals; approximately 10 minutes per assessment point): baseline, middle of the intervention, post-treatment, four-week follow-up.

INTERVENTIONS:
Behavioral: iWork.Comp — The iWork.COMP is a short-term and low-time consuming internet delivery CFT-based intervention specifically designed to mitigate the impact of toxic leadership styles through the development of compassionate motivation in the workforce of EU hospitals. The iWork.COMP encompasses 8 individual sessions (20 minutes each; mixed format including text, audio and video presentations), which will be available weekly for participants at the KEEPCARING website (https://keepcaring.eu). Each session has three parts. Part 1 encompasses a brief check-in on the stress level of the participant at that moment and on the source of their stress (if applicable). In Part 2, the theme of the session is developed. Finally, Part 3 encompasses a brief check-in on the stress level of the participant at the end of the session and on the usefulness of the session; an optional open question to provide feedback will also be displayed.
  Other Names: CFT for health care professionals
  Arms: Treatment Group

SUMMARY:
According to the literature, the prevalence of anxiety, depression, and/or burnout symptoms among healthcare workers is high. There are several factors than can, directly or indirectly, be related to these symptoms, being the leadership styles one of them. Toxic leadership, as a form of malicious leadership, has been shown to negatively impact the mental health and wellbeing of the workforce, through the adoption of dysfunctional behaviour and/or the presence of deviant personality traits (psychopathic, Machiavellianism, narcissistic) in leaders. Despite its relevance, there is an absence of studies on the efficacy of intervention programs aimed to reduce the impact of toxic leadership styles in the workplace, namely among health care professionals. Compassion Focused Therapy (CFT) is considered an effective therapeutic approach for the rehabilitation of individuals with several psychopathological symptoms/disorders (e.g., anxiety, stress, burnout, and deviant personality traits) and for the establishment of healthy relationships with friends, family, and coworkers. In the workplace, CFT-based interventions have been shown to promote employees' wellbeing, through the reduction of stress and burnout symptoms and improvement of healthy and compassionate interpersonal relationships. It is thus mandatory to develop and test cost-effectiveness CFT-based intervention programs able to mitigate the impact of toxic leadership styles in the workforce, promoting compassionate workplaces in health care systems.

To fulfil this gap, this clinical trial intends to develop and preliminarily test the efficacy of a short-term and low-time consuming internet delivery CFT-based intervention (iWork.COMP) specifically designed to mitigate the impact of toxic leadership styles through the development of compassionate motivation among health care professionals. Following a Randomized Controlled Trial, with 200 participants allocated to either a treatment group (TG) or a waiting-list control group (WLCG), it is hypothesized that the iWork.COMP will reduce the impact of toxic leadership styles, deviant traits and burnout symptoms among the TG when compared with the WLCG. Moreover, we expect that the iWork.COMP will promote wellbeing and a compassionate motivation among the TG when compared with the WLCG.

DETAILED DESCRIPTION:
1. Introduction Healthcare workers are in significant risk for the development of psychopathology, including depression, anxiety, psychological distress and burnout symptoms. According to the European Agency for Safety and Health Work (EU-OSHA; https://osha.europa.eu/en), there are several factors that may contribute to these mental health issues, such as excessive workload, conflicting demands and lack of role clarity, lack of involvement in making decisions that affect the worker, poorly managed organizational change, ineffective communication, and lack of support from management. These factors can be directly or indirectly related to leadership styles. Within leadership research, there has been an increasing interest in the study of toxic leadership, as a form of malicious leadership, in which leaders, through dysfunctional behaviour and/or deviant personality traits (psychopathic, Machiavelism, narcissistic), negatively impact on the mental health and wellbeing of the workforce. Despite its relevance, there is an absence of studies on the efficacy of intervention programs aimed at reducing the impact of toxic leadership styles in the workplace, namely among health care professionals.

   Within psychotherapeutic interventions, there has been a growing empirical support for compassion-based interventions (e.g., Compassion-Focused Therapy; CFT), in a wide range of contexts. Recent studies have shown that CFT is considered an effective therapeutic approach for the rehabilitation of individuals with several psychopathological symptoms/disorders (e.g., anxiety, stress, burnout, and deviant personality traits) and for the establishment of healthy relationships with friends, family, and coworkers. In the workplace, CFT-based interventions have been shown to promote employees' wellbeing, through the reduction of stress and burnout symptoms and improvement of healthy and compassionate interpersonal relationships. Compassion can be conceptualized as a motivation to be sensitive to the suffering of one-self and others, allied with the wisdom and commitment to prevent and/or relieve it. It is linked with psychological well-being and has been found to be negatively associated with emotion dysregulation, shame and self-criticism. In the workplace, compassion has been linked with work commitment and work satisfaction. Moreover, compassion at work has been negatively associated with burnout symptoms. It is thus mandatory to develop and test cost-effectiveness CFT-based intervention programs able to mitigate the impact of toxic leadership styles in the workforce, promoting compassionate workplaces in health care systems. These mitigation programs can impact on an individual, team, and organizational levels. Promoting a compassionate motivation among health care professionals is crucial to their mental and physical health, to their wellbeing at work, and, consequently, to the delivery of safe, high-quality, and patient-centered care to the population.
2. Study Design This study will follow a Randomized Controlled Trial design (RCT; CONSORT-Statement) involving health care units from the Health Local Unity of Coimbra (HLU Coimbra; selected by the hospital's administration). The selected health care units will be randomly assigned to the Treatment Group (TG) and to the Waiting List Control Group WLCG). The randomization at the health care unit level (and not at an individual level) intends to maximize the intervention effects, as all participants will be receiving the intervention at the same time, potentially boosting and cumulating individual and team intervention effects.

   Individuals who agree to participate in this RCT will sign an informed consent and will be asked to fulfil their socioeconomic data and a set of questionnaires (baseline assessment, M0). Participants will be assessed in three more assessment points (4-weeks intervals): middle of the intervention (M1), post treatment (M2) and 4-week follow-up (M3). All assessments (M0 to M3) will approximately take 10 minutes.
3. Participants Participants will be 200 emerging/pre-service (Gen-Z) and current health care workers (i.e., doctors and nurses working in the surgical pathway), aged over 18 years old and assuming both leader and non-leader roles in two (or more) similar Portuguese health care units. As the iWork.COMP program aims to be applied to all the workforce, no more restrictions are planned on age as well as on gender distribution.

   Regarding the sample size, a power analysis was conducted a priori (GPower v3.1 software), specifying for F tests (multivariate analysis of variances: repeated measures, within-between interaction), showing that a sample of 162 participants was necessary to detect medium effects with a significance level of .05 and a power of .90.
4. Intervention The iWork.COMP is a short-term and low-time consuming internet delivery CFT-based intervention specifically designed to mitigate the impact of toxic leadership styles through the development of compassionate motivation in the workforce of EU hospitals. The iWork.COMP encompasses 8 individual sessions (20 minutes each; mixed format including text, audio and video presentations), which will be available weekly for participants at the KEEPCARING website (https://keepcaring.eu). Each session has three parts. Part 1 encompasses a brief check-in on the stress level of the participant at that moment and on the source of their stress (if applicable). In Part 2, the theme of the session is developed. Finally, Part 3 encompasses a brief check-in on the stress level of the participant at the end of the session and on the usefulness of the session; an optional open question to provide feedback will also be displayed.

   At the end of the iWork.COMP, participants will have full access to a SOS-Button tool, which aims to provide short-term exercises when one is dealing with an acute stressful situation.
5. Measures During the four assessment moments, both TG and WLCG participants will answer a set of questionnaires already validated for the Portuguese population, aimed at measuring toxic leadership styles (Toxic Leadership Scale; TLS); deviant personality traits (Dirty Dozen; DD); burnout (Burnout Assessment Tool; BAT-12); wellbeing (Daniels's Five-Factor Measure; D-FAW), and compassion (Fears of Compassion Scales; FCS). A detailed description of these questionnaires will be presented in the outcome measures section.
6. Data analysis The data will be analyzed with SPSS v29 and Mplus v8 statistical software. Preliminary analyses, namely for comparisons between groups at baseline on sociodemographic data and outcome measures, will resort to independent-samples t-tests and chi-square tests. Internal consistency calculations will be based on Cronbach's alpha guidelines. To test the efficacy of the iWork.COMP, data will be analyzed both at an individual (Reliable Change Index) and group level (Latent Growth Curve Models). If Latent Growth Curve models don't present acceptable fit indices, treatment effects will be assessed through MANOVAs.
7. Ethical Considerations To address any ethical considerations, a series of procedures will be carried out.

First, all procedures involved in this project will be allied with the ethical principles of the Declaration of Helsinki and the European Code of Conduct for Research Integrity. Applicable national laws and regulations will also be followed. Moreover, all procedures were approved by the Ethics Committee of the Faculty of Psychology and Educational Sciences, University of Coimbra (CEDI/FPCEUC: 97/4).

Second, after the selection and randomization of the health care units, it will be conducted a series of meetings with the leaders and staff of the units. These meetings intend to inform about the nature and aims of the study, to explain the assessment procedures, to clarify any doubt that may arise, and to invite them to voluntarily participate. It will be explained that their decision to participate or not will have no negative consequences or monetary rewards, and that they can withdraw from the study at any time without further explanation. Confidentiality and anonymity will be guaranteed. Participants will fulfil a written informed consent.

Third, participants will be asked to provide their e-mail address (optional). The e-mail addresses will not be linked with the individual data of participants and will only be used to notify them regarding the availability of the sessions (for the TG) and/or assessment periods (for both TG and WLCG). Participants can ask to be removed from the mailing list at any time without further explanations.

Four, to assure data confidentiality, the following procedures will be carried out: 1) use of a system code in each research protocol; 2) unpair the research protocol and the informed consent, to maintain participants' anonymity; 3) collect personal data strictly necessary for research purposes; 4) enter data in statistical software, analyzing them exclusively in a collective way; 5) use of respondent-specific codes to link data from one time-point to the next.

Fifth, although participants in the WLCG will not receive any intervention during the study period, they will be able to access the iWork.COMP program (and then to the SOS-Button tool) after the study completion, if they choose to.

ELIGIBILITY:
Inclusion Criteria:

* Emerging/pre-service (Gen-Z) and current health care worker (i.e., doctors and nurses working in the surgical pathway);
* Aged over 18 years old;
* Assuming both leader and non-leader roles.

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
The Toxic Leadership Scale | Baseline; 4 weeks (middle intervention); 8 weeks (post-intervention); 12 weeks (Follow-up)
  Toxic Leadership: The Toxic Leadership Scale (TLS) is a 15-item instrument that aims to measure the five toxic leadership dimensions proposed by Schmidt: Abusive Supervision (i.e., the demonstration of hostile verbal and nonverbal behaviors), Authoritarian Leadership (i.e., an absolute control over his/her subordinates and all decision making), Narcissism (i.e., a grandiose and self-centered style), Self-promotion (i.e., a presentation of the self as a smart and capable person), and Unpredictability. Items are rated on a six-point Likert-type scale ranging from 1 (Strongly Disagree) to 6 (Strongly Agree). Higher total scores indicate higher levels of toxic leadership style. The TLS will be used in the present study to assess employees' perception of their direct leader's toxic leadership styles. Psychometric studies of the TLS have demonstrated a very good internal consistency (α ranging from .87 to .93).

SECONDARY OUTCOMES:
The Dirty Dozen | Baseline; 4 weeks (middle intervention); 8 weeks (post-intervention); 12 weeks (Follow-up)
  Dark Triad: The Dirty Dozen (DD) is a brief 12-item questionnaire that aims to measures the "Dark Triad", as a constellation of three overlapping, although distinct, constructs: Machiavellianism (i.e., a manipulative and cold interpersonal style), Psychopathy (i.e., a callous, unemphatic and impulsive style), and Narcissism (i.e., a grandiose and dominant style). Items are scored using a five-point Likert-type scale ranging from 1 (Totally Disagree) to 5 (Totally Agree). Higher total scores indicate higher levels of Dark Triad traits. The other-report version of the scale will be used in the present study to assess employees' perception of their direct leader's Dark Triad traits. Psychometric studies of the other-report version of the DD have demonstrated good to very good internal consistency (α ranging from .87 to .93).
The Burnout Assessment Tool | Baseline; 4 weeks (middle intervention); 8 weeks (post-intervention); 12 weeks (Follow-up)
  The Burnout Assessment Tool (BAT-12) is a brief 12-item self-report instrument that measures participant's four core burnout symptoms: Exhaustion (e.g., "At work, I feel physically exhausted."), Mental Distance (e.g., "I struggle to find any enthusiasm for my work."), Cognitive Impairment (e.g., "At work, I have problems staying focused."), and Emotional Impairment (e.g., "At work, I feel unable to control my emotions."). Items are rated on a five-point Likert-type scale ranging from 1 (Never) to 5 (Always). Higher scores indicate the participant's frequency of these symptoms. The BAT-12 will be used in the present study to assess employees' burnout symptoms and respective frequency. Psychometric studies of the BAT-12 have demonstrated good to very good internal consistency (α ranging from .85 to .95).
The Daniels's Five-Factor Measure | Baseline; 4 weeks (middle intervention); 8 weeks (post-intervention); 12 weeks (Follow-up)
  The Daniels's Five-Factor Measure (D-FAW) is a self-report questionnaire aimed at measuring participants' affective wellbeing in the past week at work. It comprised 10 items that purports to measure levels of Positive Activated Affect (PA; e.g., Happy", "At ease") and Negative Activated Affect (NA; e.g., "Anxious", "Tired"). Participants will be instructed to classify the feelings experienced using a five-point Likert-type scale ranging from 1 (Not at all) to 6 (Very much). Higher total scores indicate greater affective wellbeing at work, after the five items related to negative emotions have been reversed. Studies have demonstrated a good internal consistency for the PA and NA factors (α > .80 and .80).
The Fears of Compassion Scales | Baseline; 4 weeks (middle intervention); 8 weeks (post-intervention); 12 weeks (Follow-up)
  The Fears of Compassion Scales (FCS) include three self-report questionnaires (total of 38-items) aimed at measuring fears, blocks and resistances to the three flows of compassion as posted by the CFT framework: expressing compassion for others (10 items; e.g., "People will take advantage of me if they see me as too compassionate"); receiving compassion from others (13 items; e.g., "Wanting others to be kind to oneself is a weakness"); and being self-compassionate (15 items; e.g., "I feel that I don't deserve to be kind and forgiving to myself"). Items are rated on a five-point Likert-type scale ranging from 0 (Don't agree at all) to 4 (Completely agree). These scales have been presenting acceptable to very good internal consistencies (α ranging from .78 to .87 on the original version; ranging from .88 to .94 in the Portuguese version).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Psychology and Educational Sciences of the University of Coimbra, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hao Q, Wang D, Xie M, Tang Y, Dou Y, Zhu L, Wu Y, Dai M, Wu H, Wang Q. Prevalence and Risk Factors of Mental Health Problems Among Healthcare Workers During the COVID-19 Pandemic: A Systematic Review and Meta-Analysis. Front Psychiatry. 2021 Jun 15;12:567381. doi: 10.3389/fpsyt.2021.567381. eCollection 2021. PMID 34211406
- [Background] Batra K, Singh TP, Sharma M, Batra R, Schvaneveldt N. Investigating the Psychological Impact of COVID-19 among Healthcare Workers: A Meta-Analysis. Int J Environ Res Public Health. 2020 Dec 5;17(23):9096. doi: 10.3390/ijerph17239096. PMID 33291511
- [Background] Boucher VG, Dahl M, Lee J, Faulkner G, Beauchamp MR, Puterman E. An umbrella review and meta-analysis of 87 meta-analyses examining healthcare workers' mental health during the COVID-19 pandemic. J Affect Disord. 2025 Apr 15;375:423-436. doi: 10.1016/j.jad.2025.01.109. Epub 2025 Jan 23. PMID 39862981
- [Background] (4) LeBreton JM, Shiverdecker LK, Grimaldi EM. The dark triad and workplace behavior. Annu Rev Organ Psychol Organ Behav. 2017;5(1):387-414. https://doi.org/10.1146/annurev-orgpsych-032117-104451
- [Background] (5) Whicker ML. Toxic leaders: When organizations go bad. Quorum; 1996.
- [Background] Wasson RS, Barratt C, O'Brien WH. Effects of Mindfulness-Based Interventions on Self-compassion in Health Care Professionals: a Meta-analysis. Mindfulness (N Y). 2020;11(8):1914-1934. doi: 10.1007/s12671-020-01342-5. Epub 2020 Mar 5. PMID 32421083
- [Background] Kirby JN, Tellegen CL, Steindl SR. A Meta-Analysis of Compassion-Based Interventions: Current State of Knowledge and Future Directions. Behav Ther. 2017 Nov;48(6):778-792. doi: 10.1016/j.beth.2017.06.003. Epub 2017 Jun 21. PMID 29029675
- [Background] (9) Gilbert P, Simos G. Compassion focused therapy: Clinical practice and applications. Routledge; 2022. https://doi.org/10.4324/9781003035879
- [Background] Ribeiro da Silva D, Rijo D, Brazao N, Paulo M, Miguel R, Castilho P, Vagos P, Gilbert P, Salekin RT. The efficacy of the PSYCHOPATHY.COMP program in reducing psychopathic traits: A controlled trial with male detained youth. J Consult Clin Psychol. 2021 Jun;89(6):499-513. doi: 10.1037/ccp0000659. PMID 34264698
- [Background] Matos M, Albuquerque I, Galhardo A, Cunha M, Pedroso Lima M, Palmeira L, Petrocchi N, McEwan K, Maratos FA, Gilbert P. Nurturing compassion in schools: A randomized controlled trial of the effectiveness of a Compassionate Mind Training program for teachers. PLoS One. 2022 Mar 1;17(3):e0263480. doi: 10.1371/journal.pone.0263480. eCollection 2022. PMID 35231057
- [Background] (12) Gilbert P. Introducing compassion-focused therapy. Adv Psychiatr Treat. 2009;15(3):199-208. https://doi.org/10.1192/apt.bp.107.005264
- [Background] Zessin U, Dickhauser O, Garbade S. The Relationship Between Self-Compassion and Well-Being: A Meta-Analysis. Appl Psychol Health Well Being. 2015 Nov;7(3):340-64. doi: 10.1111/aphw.12051. Epub 2015 Aug 26. PMID 26311196
- [Background] (14) Gouveia MJ, Canavarro MC, Moreira H. Associations between mindfulness, self-compassion, difficulties in emotion regulation, and emotional eating among adolescents with overweight/obesity. J Child Fam Stud. 2018;28(1):273-285. https://doi.org/10.1007/s10826-018-1239-5
- [Background] (15) Gilbert P, Procter S. Compassionate mind training for people with high shame and self-criticism: Overview and pilot study of a group therapy approach. Clin Psychol Psychother. 2006;13(6):353-379. https://doi.org/10.1002/cpp.507
- [Background] (16) Eldor L, Shoshani A. Caring relationships in school staff: Exploring the link between compassion and teacher work engagement. Teaching and Teacher Education. 2016;59:126-136. https://doi.org/10.1016/j.tate.2016.06.001
- [Background] Buonomo I, Santoro PE, Benevene P, Borrelli I, Angelini G, Fiorilli C, Gualano MR, Moscato U. Buffering the Effects of Burnout on Healthcare Professionals' Health-The Mediating Role of Compassionate Relationships at Work in the COVID Era. Int J Environ Res Public Health. 2022 Jul 23;19(15):8966. doi: 10.3390/ijerph19158966. PMID 35897337
- [Background] Montgomery P, Grant S, Mayo-Wilson E, Macdonald G, Michie S, Hopewell S, Moher D; CONSORT-SPI Group. Reporting randomised trials of social and psychological interventions: the CONSORT-SPI 2018 Extension. Trials. 2018 Jul 31;19(1):407. doi: 10.1186/s13063-018-2733-1. PMID 30060754
- [Background] (19) Campbell JP. Behavior, Performance, and Effectiveness in the Twenty-first Century. Oxford Handbooks Online. Oxford University Press; 2012.
- [Background] Faul F, Erdfelder E, Buchner A, Lang AG. Statistical power analyses using G*Power 3.1: tests for correlation and regression analyses. Behav Res Methods. 2009 Nov;41(4):1149-60. doi: 10.3758/BRM.41.4.1149. PMID 19897823
- [Background] (21) Schmidt A. Development and validation of the Toxic Leadership Scale (master's thesis). College Park (MD): University of Maryland; 2008. Accessed from: Digital Repository at the University of Maryland. Document No.: 5358.
- [Background] (22) Mónico L, Salvador A, Santos N, Pais L, Semedo C. Lideranças Tóxica e Empoderadora: Estudo de Validação de Medidas em Amostra Portuguesa. Revista Iberoamericana de Diagnóstico y Evaluación - e Avaliação Psicológica. 2019;53(4). doi: https://doi.org/10.21865/ridep53.4.10
- [Background] Jonason PK, Webster GD. The dirty dozen: a concise measure of the dark triad. Psychol Assess. 2010 Jun;22(2):420-32. doi: 10.1037/a0019265. PMID 20528068
- [Background] (24) Antunes AL, Silva PM. Avoid the dark side: A relação entre a tríade negra da personalidade e a satisfação laboral. 2021. Available from: http:// repositorio.ispa.pt/bitstream/10400.12/8522/1/24901.pdf
- [Background] Schaufeli WB, Desart S, De Witte H. Burnout Assessment Tool (BAT)-Development, Validity, and Reliability. Int J Environ Res Public Health. 2020 Dec 18;17(24):9495. doi: 10.3390/ijerph17249495. PMID 33352940
- [Background] Sinval J, Vazquez ACS, Hutz CS, Schaufeli WB, Silva S. Burnout Assessment Tool (BAT): Validity Evidence from Brazil and Portugal. Int J Environ Res Public Health. 2022 Jan 25;19(3):1344. doi: 10.3390/ijerph19031344. PMID 35162366
- [Background] Russell E, Daniels K. Measuring affective well-being at work using short-form scales: Implications for affective structures and participant instructions. Hum Relat. 2018 Nov;71(11):1478-1507. doi: 10.1177/0018726717751034. Epub 2018 Apr 13. PMID 30270934
- [Background] (28) Valdman A. Portuguese version of D-FAW (research version). Coimbra: University of Coimbra. 2023.
- [Background] Gilbert P, McEwan K, Matos M, Rivis A. Fears of compassion: development of three self-report measures. Psychol Psychother. 2011 Sep;84(3):239-55. doi: 10.1348/147608310X526511. Epub 2011 Apr 13. PMID 22903867
- [Background] (30) Matos M, Pinto-Gouveia J, Duarte J, Simões D. The Fears of Compassion Scales. (Portuguese trans.) Unpublished manuscript. 2016.
- [Background] (31) George D, Mallery P. SPSS for Windows step by step: a simple guide and reference. 11.0 update. 4th ed. Boston (MA): Allyn & Bacon; 2003
- [Background] (32) Paulhus DL, Williams KM. The dark triad of personality: Narcissism, Machiavellianism, and psychopathy. J Res Pers. 2002;36(6):556-563. https://doi.org/10.1016/s0092-6566(02)00505-6
- [Background] (33) Mutschmann M, Hasso T, Pelster M. Dark triad managerial personality and financial reporting manipulation. J Bus Ethics. 2021;181(3):763-788. https://doi.org/10.1007/s10551-021-04959-1
- [Background] (34) Volmer J, Koch IK, Göritz AS. The bright and dark sides of leaders' dark triad traits: Effects on subordinates' career success and well-being. Pers Individ Dif. 2016;101:413-418. https://doi.org/10.1016/j.paid.2016.06.046